CLINICAL TRIAL: NCT04176614
Title: Functional Cereal-based Products Fortified With Legumes for Satiety and Weight Management
Brief Title: Cereal-based Products Fortified With Legumes and Effects on Body Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Amalia Yanni, Research and Teaching Associate-Staff, Principal Investigator, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 62/03072018
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Overweight and Obesity
Keywords: cereal-based snack fortified with legumes; body weight reduction
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Overweight/obese non diabetic subjects will follow an energy-restricted diet and supplemented with a cereal-based snack fortified with legumes (intervention group) or a common cereal snack (control group) for 12 weeks. Body weight, anthropometric, clinical and biochemical characteristics will be evaluated at the beginning and at the end of the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cereal-legume snack (Experimental): Certain amount of cereal-legume snack daily for 12 weeks
  Interventions: Other: cereal-legume snack
- cereal snack (Active Comparator): Certain amount of cereal snack daily for 12 weeks
  Interventions: Other: cereal snack

INTERVENTIONS:
Other: cereal-legume snack — cereal-legume biscuit
  Arms: cereal-legume snack
Other: cereal snack — cereal biscuit
  Arms: cereal snack

SUMMARY:
Legumes are high nutritional quality foods and constitute a rich source of proteins and dietary fibers which have been associated with appetite regulation and body weight management. The purpose of the study is to investigate the effects of regular consumption of a cereal-based snack fortified with legumes on body weight reduction.

DETAILED DESCRIPTION:
Overweight/obese, non-diabetic subjects will participate in the study. Subjects will follow a 12-week energy-restricted dietary intervention supplemented with a certain amount of a cereal-based snack fortified with legumes daily. The effects of dietary intervention on body weight reduction will be examined.

ELIGIBILITY:
Inclusion Criteria:

* normal exercise and dietary habits
* weight stable for at least 3 months before enrollment

Exclusion Criteria:

* diabetes
* pregnancy
* chronic medical illness
* use of nutritional supplements
* regular intense exercise
* alcohol consumption > 2 drinks/day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 12 weeks
  Change in body weight after energy-restricted dietary intervention with cereal-legume snack compared to common cereal snack

CONTACTS AND LOCATIONS:
Overall Officials: Amalia Yanni, Dr, Principal Investigator — Harokopio University; Alexander Kokkinos, Prof, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Laiko General Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No